CLINICAL TRIAL: NCT01446978
Title: Hepatitis A Vaccination in Patients With Rheumatoid Arthritis Treated With TNF-inhibitors and/or Methotrexate
Brief Title: Three Doses of Hepatitis A Vaccine in Patients With Immunomodulating Drugs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Lars Rombo, Professor, Sormland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rombo - 2
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Vaccine Response Impaired
Keywords: hepatitis A vaccine; TNF-alfa inhibitory drugs; Rheumatoid arthritis; methotrexate
MeSH Terms: conditions — Hepatitis; Arthritis, Rheumatoid | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- initial single dose of hep A vaccine (Active Comparator): The participants will receive a single dose of hepatitis A vaccine at 0+1+6 months
  Interventions: Biological: hepatitis A vaccine
- initial double dose (Active Comparator): Participants will receive one dose of hepatitis A vaccine in each M. deltoids and an additional dose at 6 months later
  Interventions: Biological: hepatitis A vaccine

INTERVENTIONS:
Biological: hepatitis A vaccine — 3 doses of hepatitis A vaccine, given at 0+1+6 months
  Arms: initial single dose of hep A vaccine
Biological: hepatitis A vaccine — Two doses of hepatitis A vaccine given at day 0, one in each M deltoids. An additional dose will be given at 6 months later
  Arms: initial double dose

SUMMARY:
Hepatitis A vaccine is the most frequently used traveler's vaccine, yet data on its ability to induce protective immunity in immunosuppressed travelers are scarce. The investigators assess the hepatitis A virus (HAV) antibody response in patients with rheumatoid arthritis (RA) treated with Tumor Necrosis Factor (TNF) - inhibitors and/or methotrexate (Mtx).

In a previous study, 2 doses were not considered effective and there is therefore need for a study with an additional dose

DETAILED DESCRIPTION:
Methods: Parameters registered at baseline were: age, sex, duration of disease, medications, activity of disease (Visual Analogue Scale), Health Assessment Questionnaire Disability Index, Disease Activity Score, Acute phase reactant and total immunoglobulin G in plasma). Hepatitis A vaccine (Epaxal or Havrix) were given at 0 and 6 months. Hepatitis A virus (HAV) antibodies is measured before vaccination and at month 1, 6 (before dose 2), 7 and 12 with quantitative HAV IgG, using the HAVAb-IgG Architect System, and by the HAVAB 2.0 assay on the AxSYM machine from Abbott. The level of protective immunity to HAV is defined as HAV IgG > 10mIU/mL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis
* TNF-alfa blocker and / or methotrexate in use as a medication against RA
* A desire to get protected against hepatitis A
* Men and women age 18-65 years
* Written informed consent
* Women of childbearing potential must use effective contraception -

Exclusion Criteria:

* Treatment with rituximab within 9 months before study start
* Known previous hepatitis A infection
* Previous vaccination against hepatitis A
* Allergy to eggs or formaldehyde
* Pregnancy or lactation
* Excessive use of alcohol
* Mental retardation
* Acute disease at the time of examination (fever > 38 degrees)
* Volunteer works as an employee of the researchers
* Previous vaccination against hepatitis A
* Egg-, hen-protein- or formaldehyde allergy
* Pregnancy or lactation
* Excessive use of alcohol
* Another vaccine given within a month
* Acute disease at the time of examination (fever > 38 degrees)
* Not suitable for other reason in the investigator's opinion (other serious disease, i.e. AIDS/HIV-positive, cancer with ongoing cytostatic treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
seroconversion after the first dose/doses of hepatitis A vaccine | one month after the first dose/doses
  ELISA-titers are determined before the first dose/doses and at 1 month later

SECONDARY OUTCOMES:
seroconversion rates after three doses of hepatitis A vaccine | 12 months after the first doses
  We determine seroconversion rates before the third vaccine dose (6 months after the first) and at 1 and 6 months after the second dose

CONTACTS AND LOCATIONS:
Overall Officials: lars rombo, MD, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Dept infectious diseases, Eskilstuna
  - Dept infectious diseases, Örebro
  - Department of infectious diseases, Stockholm
  - Dept infectious diseases, Uppsala